CLINICAL TRIAL: NCT01206660
Title: A Double-Blind, Vehicle-Controlled, Randomized, Parallel Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone 0.25% Topical Spray in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Effects of Desoximetasone Spray 0.25% in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSXS-0914
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desoximetasone Spray 0.25% (Experimental): Desoximetasone topical spray 0.25% administered to affected area twice a day for 28 days
  Interventions: Drug: Desoximetasone Spray 0.25%
- placebo (Placebo Comparator): Placebo administered to affected area twice a day for 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Desoximetasone Spray 0.25% — Desoximetasone topical spray 0.25% administered to affected area twice a day for 28 days
  Arms: Desoximetasone Spray 0.25%
Drug: placebo — Placebo administered to affected area twice a day for 28 days
  Arms: placebo

SUMMARY:
The objective of this study is to demonstrate that desoximetasone 0.25% topical spray is effective for the treatment of patients with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 18 years of age or older.
* Have a definite clinical diagnosis of stable plaque psoriasis involving ≥ 10% of the body surface area (BSA).
* Have a combined total lesion severity score (TLSS) of ≥ 7 for the Target Lesion.
* Have a plaque elevation score ≥ 3 of (moderate) for the Target Lesion.
* The Target Lesion must have an area of at least 5 cm².
* Have a Physicians Global Assessment (PGA) score of 3 (moderate) or 4 (severe) at baseline for the overall disease severity.

Exclusion Criteria:

* Patient has current diagnosis of other types of psoriasis other than stable plaque psoriasis (i.e. acute, guttate, erythrodermic, exfoliative or pustular psoriasis) or has psoriasis of any kind of the face or scalp that will require active treatment during the study. Nonprescription antipsoriatic shampoos will be allowed during the study when applied solely to the scalp.
* Patient has a history of psoriasis that has been unresponsive to topical corticosteroid therapy.
* In the Investigator's opinion, the patient has other dermatological conditions, such as atopic or contact dermatitis, that may interfere with the clinical assessments of the signs and symptoms of psoriasis.
* Patient has a history of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
* Patient has been treated within 12 weeks (or five half lives, whichever is less) prior to the first dose of study drug with any biological therapies for psoriasis.
* Patient has received any systemic steroids within 4 weeks of the first dose of the study drug. The use of inhaled or intranasal corticosteroids is acceptable as long as usage has been stable for at least 2 weeks prior to the first dose of study drug and will be continued during the study.
* Patients who have used any topical antipsoriatic agents of any kind or any topical corticosteroids for any reason within 2 weeks prior to first use of study drug. Nonprescription antipsoriatic shampoos used only on the scalp will be allowed during the study.
* Receipt of any drug as part of a research study within 30 days prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site, Hazleton, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desoximetasone Spray 0.25% | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.03 (14.29) | 53.55 (14.82) | 50.79 (14.56)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 13 | 30
  Between 18 and 65 years | 34 | 31 | 65
  >=65 years | 9 | 16 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 37 | 35 | 72
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success ITT
Description: A patient is considered a Clinical Success if the Physician's Global Assessment (PGA) is 0 (clear) or 1 (almost clear).
Time Frame: 28 days
Population: Analysis was conducted using Intent-to-Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 60 | 60
participants | 32 | 11
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Treatment Success
Description: A patient is considered a Treatment Success for the Target Lesions if the target lesion has a score of 0 or 1 on the Target Lesion Severity Score (TLSS) for each the three signs and symptoms (erythema, scaling and plaque elevation).
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 60 | 60
participants | 32 | 10
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Physician's Global Assessment (PGA) of Psoriasis Score at Day 28.
Description: Physician Global Assessment (PGA) of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of face, genitals, or intertriginous area (i.e., breast fold, gluteal crease, axilla). Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease.
Time Frame: Day 28
Population: ITT Population. Participants who returned for at least one post baseline visit and/or provided an assessment for pruritus were evaluated; not all participants returned for every study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 60 | 60
units on a scale | 1.73 (1.06) | 0.85 (0.94)
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 4/60 | 5/60
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desoximetasone Spray 0.25% (N=60) | Placebo (N=60)
Application Site Irritation (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
Application Site Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No